CLINICAL TRIAL: NCT03801395
Title: Primary Ciliary Dyskinesia New Gene Discovery to Improve Diagnostics and Clinical Care
Brief Title: PCD New Gene Discovery
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Michael O'Connor, Assistant Professor, Vanderbilt University Medical Center
Other Study IDs: 182074
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Primary Ciliary Dyskinesia
MeSH Terms: conditions — Ciliary Motility Disorders

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be obtained for DNA analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: There is no intervention — No intervention

SUMMARY:
This is a new gene discovery program for individuals with PCD who do not have a specific genetic etiology identified. Research procedures involve a single blood draw from the affected individual and from unaffected family members in an effort to identify new genetic targets.

DETAILED DESCRIPTION:
The objective of this study is to better define how the genes that cause primary ciliary dyskinesia (PCD) are related to the clinical symptoms of individuals with PCD. PCD is a rare disease that affects the function of motor cilia throughout the body. This results in a variety of clinical symptoms, but chief among them are a chronic wet cough, recurrent sinusitis, and frequent pneumonia. These clinical symptoms can result in further structural lung disease, including bronchiectasis, with eventual worsening of lung function. The treatment for this condition largely focuses on augmenting airway clearance and appropriate use of antimicrobial therapies, in conjunction with monitoring for evidence of pulmonary impairment. Thus, it is important to identify and diagnose individuals with PCD early in life.

Making a diagnosis of PCD can be difficult as their is some overlap of the clinical symptoms with other conditions and there are limitation in the current diagnostic testing modalities. Historically, the diagnosis has been made by identification of structural abnormalities in cilia by electron microscopy (ciliary biopsy). However, this testing has limitations secondary to the somewhat invasive nature of the procedures and often inconclusive results secondary to sampling challenges (getting enough cilia). Furthermore, a normal ciliary biopsy result does not rule-out PCD as it is now known that there are individuals with PCD who have ciliary dysfunction secondary to ciliary abnormalities that are not routinely identified on standard electron micrograph. Genetic testing for PCD is available, but current testing only accounts for about 60-65% of the PCD population. Thus normal results in this regard do not rule-out PCD either. Nasal nitric oxide (nNO) testing is an emerging research-based testing that is being used more frequently to identify individuals with PCD. More specifically, it has been frequently observed that individuals with PCD have low levels of nitric oxide in their sinus cavities. Measuring a low level of nitric oxide of multiple different occasions has proven to have diagnostic utility in an individual with a clinical symptom history consistent with PCD. While nNO testing is helpful for identifying individuals likely to have PCD, this testing does not give further information as to reason for ciliary dysfunction. Current testing availability has resulted in a group of individuals who are being managed as "probable PCD" which is defined by having clinical symptoms consistent with PCD (such as year-round wet cough and rhinitis) at least two separate positive (low value) nNO testing results, but negative PCD genetics and a non diagnostic ciliary biopsy. While these individuals are often managed the same as other individuals with more defined PCD, including augmentation of airway clearance therapies, in order for more specific care to be applied in the future it is important to better define the ciliary structural reason for their clinical symptoms. This could also be described as needing to better understand the genotype-phenotype of all individuals with PCD.

This investigation seeks to better define the genotypic-phenotypic relationship of individuals by initially focusing on new gene discovery in individuals with probable PCD. More specifically, through whole-exome evaluation of individuals with probable PCD and unaffected first-degree relatives, we will focus on identifying new mutations in ciliary structural proteins and other related pulmonary genes. New gene targets will then be further studied through analysis of ciliary structure and function.

ELIGIBILITY:
Inclusion Criteria:

* • Age 0-90 years

  * Confirmed diagnosis of PCD by either ciliary ultrastructure abnormality or two known disease-causing alleles in a known PCD gene OR individuals with clinical suspicion of PCD without a confirmatory test (genetics or ciliary biopsy) as defined by: low nasal nitric oxide testing (<77nl/min) on two separate occasions at least two months apart or compatible clinical phenotype, but unable to do nasal nitric oxide testing secondary to age or other factors OR relative of one of the previously defined individuals with PCD
  * Ability to provide informed consent or consent of parent/guardian and assent for minors

Exclusion Criteria:

* • Inability to understand the requirements of the study or be unwilling to provide written informed consent (as evidenced by signature on an informed consent document approved by the IRB) OR inability of parent/guardian to understand the requirements of the study

Ages: 0 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with confirmed or suspected PCD and their unaffected family members
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
DNA analysis | 6 months
  Blood will be obtained for DNA analysis and identification of new PCD genes. Genetic analysis will be done by whole exome sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt Children's hospital, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No